CLINICAL TRIAL: NCT04299386
Title: A Randomized Clinical Trial on the Effect of Nanocrystal Gels on the Management of Peri-implant Diseases
Brief Title: Effect of Nanocrystal Gels on the Management of Peri-implant Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Robert Durand, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CERC-19-084-P
Record Dates: First submitted 2020-03-01; First posted 2020-03-06 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Dental Implant Failure Nos
Keywords: Dental implants; Infection control; Bone Healing; professional cleaning

STUDY DESIGN:
Intervention Model Description: Double-masked parallel-arm randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NeoPhylaxis (Experimental): Nanocrystalline gel for nonsurgical cleaning of implants
  Interventions: Device: NeoPhylaxis
- ImplanTreat (Experimental): Nanocrystalline gel for surgical cleaning of Implants
  Interventions: Device: ImplanTreat
- Nonsurgical cleaning without gel (No Intervention): Cleaning dental implants non-surgically using the electric brush without the gel
- Surgical cleaning without gel (No Intervention): Cleaning dental implants surgically using the electric brush without the gel

INTERVENTIONS:
Device: NeoPhylaxis — NeoPhylaxis® gel is designed for the non-surgical decontamination of the implant surface and can be used for professional regular implant maintenance, with or without peri-implant mucositis. It contains the same ingredients, Magnesium Phosphate (3.02% w/v) and Sodium Phosphate (8.23% w/v) in 3 mL syringe in non-sterile form.
  Arms: NeoPhylaxis
Device: ImplanTreat — ImplanTreat® gel can be used for the surgical decontamination of the implant surface and can be used to decontaminate implants with peri-implantitis. It contains the same ingredients, Magnesium Phosphate (3.02% w/v) and Sodium Phosphate (8.23% w/v) in 3 mL syringe in sterile form.
  Arms: ImplanTreat

SUMMARY:
Dental implants are a well-accepted treatment for replacing missing teeth, due to excellent patient satisfaction regarding function, aesthetics, and comfort, as well as their long-term survival. However, the accumulation of bacterial biofilm on implants changes their surface biocompatibility and initiates peri-implant diseases, such as peri-implant mucositis and peri-implantitis. Professional cleaning of the implant surface is necessary to remove the biofilm and facilitate healing within the surrounding tissue. Prophylaxis pastes can be used in dental clinics to assist the mechanical removal of biofilm by dental professionals. However, these pastes can contain abrasives that detrimentally affect the surface stability and chemical properties of the implant surfaces.

ImplanTreat® and Neophylaxis® are novel nanocrystal gels designed for implants' professional cleaning, under surgical and non-surgical procedures respectively. These products present high biocompatibility proprieties that can improve peri-implant bone healing. Moreover, they don't contain abrasives, or fluoride, which preserves the implant surfaces. The researchers hypothesize that professional implant cleaning with Neophylaxis® or ImplanTreat® results in a greater reduction of peri-implant inflammation and dental plaque accumulation in comparison to cleaning without any product. Accordingly, the purpose of this study is to verify if Neophylaxis® and ImplanTreat® enhance the efficacy of professional cleaning and preserve implant surface roughness.

The researchers will randomly divide the recruited participant into two groups depending on the clinical diagnosis, each patient will be either recruited in peri-implant mucositis group (Group I), or in peri-implantitis group (Group II). Each patient in the group I will be assigned randomly to receive either implant cleaning with Neophylaxis® or cleaning without. Similarly, each patient in group II will be assigned randomly to receive either implant cleaning with ImplanTreat® or cleaning without. No participant will be aware of his allocation before the end of data collection. In each evaluation session, The researchers will examine the participants' implants and evaluate the removal of biofilm as well as the improvement of the peri-implant tissue health and bone level. The researchers will then analyze and compare the results obtained from each study group.

DETAILED DESCRIPTION:
Background:

Oral hygiene and regular maintenance are crucial to sustaining healthy peri-implant tissues. However, current available prophylaxis products and toothpaste tend to contaminate and abrade the surface of implants, due to the high affinity of humectants, thickeners and surfactants to the implant surface and the high abrasiveness of silica microparticles used in these products. Nanocrystalline magnesium phosphate (NMP) gel, a novel inorganic colloidal suspension, is the result of 7 years of research in Dr. Faleh Tamimi's laboratory in collaboration with researchers from McGill University. It is a hydrogel with unique biocompatibility that can improve peri-implant bone healing. The NMP gel forms highly stable inorganic colloidal suspensions with interesting rheological properties (i.e. thixotropy) that are ideal for toothpaste and prophylaxis paste applications and do not require the addition of organic thickeners. The product contains magnesium phosphate (3.02% w/v) and sodium phosphate (8.23% w/v) in 3 mL syringe.

Hypotheses (null):

Professional cleaning of implant surfaces with NMP prophylactic gel during maintenance visits will result in similar reductions of gum redness, bleeding and plaque scores after 4 weeks than implant surfaces cleaned without gel.

Professional cleaning with NMP treatment gel of implant surfaces diagnosed with peri-implantitis will result in similar reductions of peri-implant probing depth, bleeding, plaque scores and suppuration after 4 weeks, as well as improved bone levels after 6 months, compared to implant surfaces, cleaned without gel.

Objectives:

To assess if professional cleaning of dental implants and abutments with signs of mucositis using NMP gel, during maintenance visits has better outcomes when compared to the cleaning without gel.

To assess if professional cleaning of dental implants and abutments with the NMP treatment gel, is more efficient in controlling the infection around implants with peri-implantitis than cleaning without gel.

Study design: This study will be conducted as a prospective, randomized controlled trial. The study is categorized as pivotal study and is intended to collect clinical evidence on the efficacy and safety of the tested product in a statistically justified number of subjects based on FDA classification of clinical trials for medical devices; it is equivalent to a Phase 3 clinical trial in the classification scheme for clinical trials of pharma products. The intervention group will receive the professional dental implant and abutment cleanings with NMP gel after flap elevation surgery and irrigation (ImplanTreat®, Invicare, Montreal, Canada), while the control group will receive also flap elevation surgery with irrigation but without gel application.

The participants' recruitment will take place at the implantology dental clinic of the 3 participating universities: McGill University (Montreal, QC), Université de Montréal (Montreal, QC), and Harvard University (Boston, US). Potential study participants will be identified from populations of implant-supported/retained prosthesis wearers: patients with removable and/or fixed implant- prosthesis who visit the mentioned clinics during the period of study recruitment. During their visit to the dental clinic, patients will receive an oral, periodontal and radiographic examination. Intraoral photographs will be taken at baseline for all the participants to confirm the diagnoses of peri-implantitis. Patients will be invited to participate in the trial if the oral examination confirms a diagnosis of peri-implantitis, defined as bleeding/suppuration after probing on at least one peri-implant site (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual aspects), combined with peri-implant bone loss ≥ 3 mm and probing depth ≥ 6 mm[46], justifying a surgical treatment. In the case of patients with two or more implants that show peri-implantitis, only one implant per patient will be randomly allocated into an intervention or control group. All patients meeting eligibility criteria will meet with the study coordinator and will have to sign consent forms if they are interested.

To be considered for inclusion in the study, patients should meet the following criteria:

Male or female patients aged 18 years and older. Patients with upper or lower implant-supported/retained prostheses. The implant should be in function for 12 months or more. To be included in group I, peri-implant mucositis should be diagnosed. To be included in group II, peri-implantitis should be diagnosed.

Patients will be excluded from participating in the study if they meet these exclusion criteria:

Patients who have undergone radiotherapy in the head and neck region, chemotherapy or systemic long-term corticosteroid treatment; Patients receiving medications known to induce gingival hyperplasia; Patients who have taken systemic antibiotics less than 3 months prior to baseline; Patients with prosthetic factors that prevent clinical measurements Implants with technical complications, such as poor marginal contour or any type of prosthetic complication that would be a local contributing factor to chronic inflammation.

Peri-implant bone loss > 50% [47] Presence of any acute oral infection. Presence of uncontrolled diabetes or other systemic diseases. Intravenous bisphosphonates Oral bisphosphonate intake for more than 3 years. Both cleaning procedures, with and without NMP gel, will be provided by the same dental professional. Measurements will be performed at baseline and at follow up visits by a second blinded dental professional. Data will also be analyzed by a statistician who will be blinded to the intervention assignment. Participants will also be blinded during the study intervention and follow-up.

A research assistant will be responsible for the coding process and giving the coded data to the biostatistician. The coding for the trial arms will be withheld from the examiners until data analysis is complete.

Remove the screw-retained bridge or removable prosthesis. The intervention group will receive the professional dental implant and abutment cleanings with NMP gels (NeoPhylaxis® or ImplanTreat®), while the control group will receive the professional dental implant and abutment cleanings without gel.

Participants will be classified into 2 groups, based on their peri-implant clinical condition, to separately answer the two main objectives of the trial. Group, I will include patients with peri-implant mucositis, and group II will include patients with peri-implantitis. Participants in group I will then be randomized to either NeoPhylaxis® or control, and participants in group II will be randomized to either ImplanTreat® or control.

The intervention group will receive the professional dental implant and abutment cleanings with NMP gels (NeoPhylaxis® or ImplanTreat®), while the control group will receive the professional dental implant and abutment cleanings without gel. Participants will be classified into 2 groups, based on their peri-implant clinical condition, to separately answer the two main objectives of the trial. Group, I will include patients with peri-implant mucositis, and group II will include patients with peri-implantitis. Participants in group I will then be randomized to either NeoPhylaxis® or control, and participants in group II will be randomized to either ImplanTreat® or control.

Group I cleaning procedure: For participants allocated to NMP gel only, apply NeoPhylaxis® gel on the implant/abutment surface and on the rotary brush. For the control group, cleaning will be done with the rotary brush alone and no gel will be applied. The rotary brush will be held perpendicularly while gently touching the contaminated implant surface and moving at a circular motion speed of ~2,500 rpm for ~20 seconds. The surface will be brushed thoroughly until all visual contaminants are removed, followed by water irrigation to remove contaminants and any remaining gel.

Group II cleaning procedure: Proceed with local anesthesia, then supra-crestal incision, full-thickness mucoperiosteal flap elevation; granulation tissue removal using Teflon curettes and irrigation with sterile saline (Gracey; Hu-Friedy) [48].For participants allocated to NMP gel, apply ImplanTreat® gel on the implant/abutment surface and on the rotary brush that will move at a speed of 2,500 rpm for ~20 seconds. For the control group, no gel will be applied. The surface will be brushed thoroughly until all visual contaminants are removed, followed by water irrigation to remove contaminants and any remaining gel.

Postoperative follow-up will take place after 2 weeks. During the first 2 weeks after surgery, no oral home care should be done by the participants. Thereafter, participants will be told to resume routine oral hygiene. Data will be collected in a blinded fashion by a trained and calibrated dental professional (dentist or dental hygienist) using study questionnaires, a clinical form, and standardized radiographs (using an occlusion jig material). Follow-up data collection will be performed at 4 weeks and at 6 months by the same examiner at each research center. Since this is a multicenter clinical trial, and in order to avoid bias in data collection and measurements, the PI (or Co-PI) will visit each center to train and calibrate collaborators in the other centers. Standardization will concern all study procedures, from screening potential participants to data collection and measurements. In addition, regular meetings (in person or video calls) between the PI (or Co-PI) and the principal collaborator in each center will be planned to ensure the trial follow-up.

Clinical and radiographic assessment: To assess the potential efficacy of NMP gel, outcomes include clinical and radiological measurements. Periodontal examination at 6 sites around each included implant (mesiobuccal, buccal, distobuccal, mesiolingual/ palatal, lingual and distolingual/palatal) will be performed to record the clinical periodontal indices and for every clinical index, a mean value will be calculated based on the average of the obtained values in the 6 examined sites around the implant. The primary outcome will be probing depth (PD), which will be measured in millimeters around the implant, using a UNC15 periodontal probe. Other secondary outcomes will be:

Modified Gingival Index (MGI) in which the gingivae are given a score on a five-point scale from 0 (absence of inﬂammation) to 4 (severe inﬂammation) [49].

Modified plaque index (mPI) will be recorded by running the periodontal probe across the marginal surface of the implant and recording either the absence or the presence of plaque as follows: A score of 0 represents no plaque, 1 represents separate flecks of plaque at the cervical margin; 2 represents plaque can be seen by naked eye, 3 represents abundance of soft matter.

Bleeding on probing (BoP) will be recorded using a 3-graded index 10s after probing as follows: A score of 0 represents no bleeding, 1 represents isolated minimal bleeding spots, 2 represents blood forming a confluent red line on the margin and 3 represents heavy or profuse bleeding.

Suppuration (Sup) will be evaluated by assessing the presence or absence of suppuration up to 15 seconds after probing.

Radiographic crestal bone level (CBL) will be measured on the intraoral periapical radiographs at baseline and at 6 months follow-up to assess the effect of ImplanTreat® on peri-implant bone remodeling. CBL will be measured by the distance from the implant/abutment interface to the first bone-to-implant contact on both the mesial and distal implant side. CBL will be recorded by calculating the average distances between the mesial and distal sides[48]. In order to avoid any bias, one investigator, blinded to the treatment group, will use the same X-ray device, with the same settings, for pre- and post-intervention radiographs, following a standardized procedure.

Descriptive analysis will be performed on the sociodemographic and explanatory variables. The normality of the distribution of the primary outcomes data will be initially tested. T-test and a repeated measure analysis of variance (ANOVA) will be used to compare the mean differences in the continuous variables from baseline to 4 weeks and 6 months post-intervention, between the group who received the gel cleaning with ImplanTreat® and the controls. In the case of non-normal data distributions, the Mann-Whitney and Friedman tests will be used instead of the t-test and ANOVA, respectively. P values will be considered as statistically significant if less than 0.05.

The primary outcome for the group I is the absence of bleeding on probing (BoP). Considering a clinically relevant difference of 20% in terms of frequency in BoP-positive sites between the two study groups at the 4-week follow-up, a sample size of 100 patients per treatment group has 80% power to detect a significant difference (α = 0.05) based on variability data from Lerario et al. (2016)[52]. To compensate for possible dropouts, the sample size will be increased by 10%, requiring 220 patients; including 110 test participants and 110 controls. The sample size has been calculated for Group II using PD as the primary outcome (Power and Sample Size Calculations Software, Version 3.0, Vanderbilt University, Nashville, TN, USA). In order to detect a 40% difference in terms of PD reduction between groups after 6 months with a p-value of 0.05 and 85% statistical power a sample of 154 participants will be required (77 participants per group) (Schwarz F et al 2013). The researchers anticipate an attrition rate of 10%. Consequently, 170 participants including 85 test participants and 85 controls.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years and older.
* Patients with upper or lower implant-supported/retained prostheses.
* The implant should be in function for 12 months or more.
* To be included in group I, peri-implant mucositis should be diagnosed.
* To be included in group II, peri-implantitis should be diagnosed.

Exclusion Criteria:

* Patients who have undergone radiotherapy in the head and neck region, chemotherapy or systemic long-term corticosteroid treatment;
* Patients receiving medications known to induce gingival hyperplasia;
* Patients who have taken systemic antibiotics less than 3 months prior to baseline;
* Patients with prosthetic factors that prevent clinical measurements
* Implants with technical complications, such as poor marginal contour or any type of prosthetic complication that would be a local contributing factor to chronic inflammation.
* Peri-implant bone loss 50% [47]
* Presence of any acute oral infection.
* Presence of uncontrolled diabetes or other systemic diseases.
* Intravenous bisphosphonates
* Oral bisphosphonate intake for more than 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Bleeding on probing index | 4 weeks, 6 months, 1 year
  semi-quantitative assessment of bleeding after probing around each implant 0 = No bleeding
  1. Isolated minimal bleeding spots
  2. Blood forming a confluent red line on the margin
  3. Heavy or profuse bleeding
Change in Probing depth (PD) | 4 weeks, 6 months, 1 year
  probing depth in mm of peri-implant tissues around each implant

SECONDARY OUTCOMES:
Modified Gingival Index | 4 weeks, 6 months, 1 year
  semi-quantitative assessment of gingival health around each implant 0 Absence of inflammation;
  1. Mild inflammation or with slight changes in color and texture but not in all portions of gingival marginal or papillary
  2. Mild inflammation, such as the preceding criteria, in all portions of gingival marginal or papillary
  3. Moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary
  4. Severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration
modified plaque index | 4 weeks, 6 months, 1 year
  semi-quantitative assessment of plaque around each implant(1 = Plaque only detected by running a probe along the smooth surface of the healing abutment, 2 = Plaque can be seen by the naked eye, 3 = Abundance of soft matter)
gingival suppuration after probing | 4 weeks, 6 months, 1 year
  presence or absence of pus exudate after probing around each implant
Crestal bone level (CBL) | 6 months, 1 year
  variations in mm of the alveolar bone around each implant

CONTACTS AND LOCATIONS:
Overall Officials: Robert Durand, Principal Investigator — Université de Montréal